CLINICAL TRIAL: NCT04402736
Title: Feasibility and Effectiveness of a Modified Barthel Index-based Rehabilitation Nursing Program for Acute Ischemic Stroke
Brief Title: Feasibility and Effectiveness of Rehabilitation Nursing for Acute Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018LS112
Record Dates: First submitted 2020-05-16; First posted 2020-05-27 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-05

CONDITIONS: Acute Ischemic Stroke; Nursing
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Barthel Index-based rehabilitation nursing program (Experimental): Patients received the Modified Barthel Index based rehabilitation nursing from qualified nurses.
  Interventions: Behavioral: The modified Barthel Index-based rehabilitation nursing program
- Usual care (Other): Patients received the usual care.
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: The modified Barthel Index-based rehabilitation nursing program — The intervention with the program based on the MBI classified function of patients into five levels, with every 20 points as a level, Each level corresponds to different training items. Training items included self-care training and training in transfer activities, sitting balance, walking, and sit-to-stand, etc. Each training session lasting at least 30 minutes, two sessions per day, for seven continuous days. During the intervention, the rehabilitation therapist's conventional treatment is not interfered.
  Arms: Modified Barthel Index-based rehabilitation nursing program
Behavioral: Usual care — Patients in the control group received clinical usual care including the activities of daily living assessment, early mobilization guide and health education. During the intervention, the rehabilitation therapist's conventional treatment is not interfered.
  Arms: Usual care

SUMMARY:
In the clinical setting, it is difficult to obtain effective rehabilitation during the acute phase, the reasons may include insufficient awareness of early rehabilitation due mainly to a limitation in number and variety of rehabilitation professionals in Low- and middle-income countries. It is necessary to shift tasks to other healthcare providers who are trained to provide rehabilitation like nurses. The purpose of this study is to examine the feasibility and effectiveness of a modified Barthel Index based rehabilitation nursing program on acute stroke inpatients.

DETAILED DESCRIPTION:
Ischemic stroke is the main cause of disability in the world. More than 70% of stroke patients show various degrees of neural function impairment. Early rehabilitation in acute phase is beneficial for improving patient's activity of daily livings and motor function. However, it is difficult to obtain effective rehabilitation during the acute phase of stroke because of the insufficiency of professional rehabilitation therapists in stroke wards in China. The investigators assume that implementing program based on modified Barthel Index can realize nursing-directed motor rehabilitation during acute phase of ischemic stroke. The present study is to conduct quasi-experimental research to confirm the feasibility and effectiveness of nursing-directed precision rehabilitation in acute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with ischemic stroke and met the diagnostic criteria of the World Health Organization;
* initial stroke within seven days, with limb dysfunction;
* NIHSS scale consciousness scores of 0 or 1;
* provided informed consent form.

Exclusion Criteria:

* incomplete clinical data;
* having a physical disability or other diseases that affect the limb function;
* having cognitive impairment or other diseases that interfere with participation;
* having serious cardiopulmonary dysfunction or another disease that requires absolute bed rest;
* having progressive stroke or having severe complications that patients drop the study before completion.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline the Modified Barthel Index (MBI) on day 7 | Day 0 and day 7
  The MBI score ranges from 0 to 100, the higher scores mean a better outcome.
Change from baseline the motor assessment scale (MAS) on day 7 | Day 0 and day 7
  The MAS scale excluding general tonus, may be summed to provide an overall score out of a possible 48 points and the higher scores mean a better outcome.
Change from baseline the National Institute of Health Stroke Scale (NIHSS) on day 7 | Day 0 and day 7
  The NIHSS scale ranges from 0 to 42, and the higher scores mean a worse outcome.

SECONDARY OUTCOMES:
The completion rate | Day 7
  The completion means participants completed all the study stage and all the data collection.
The adverse events rate | Day 7
  The adverse events including pneumonia, stroke progression or recurrent, fall.

CONTACTS AND LOCATIONS:
Overall Officials: Jingfen Jin, Master, Study Director — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China